CLINICAL TRIAL: NCT03867318
Title: A Phase III Double-Blind Efficacy and Safety of Ezetimibe (SCH 58235) 10 MG in Addition to Atorvastatin in Subjects With Coronary Heart Disease or Multiple Cardiovascular Risk Factors and With Primary Hypercholesterolemia Not Controlled by a Starting Dose (10 mg) of Atorvastatin
Brief Title: Efficacy and Safety Study of Ezetimibe (SCH 58235, MK-0653) in Addition to Atorvastatin in Participants With Coronary Heart Disease or Multiple Cardiovascular Risk Factors (P00693/MK-0653-030)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P00693; MK-0653-030 (Other: Merck Protocol Number); P00693 (Other: Schering Plough Protocol Number)
Record Dates: First submitted 2019-03-06; First posted 2019-03-07 (Actual); Last update posted 2024-05-10 (Actual); Status verified 2022-02

CONDITIONS: Hypercholesterolemia
MeSH Terms: conditions — Hypercholesterolemia | interventions — Atorvastatin; Ezetimibe

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Atorvastatin Monotherapy (Experimental): Participants receive double-blind atorvastatin 10 mg once daily (QD) via oral tablet PLUS open-label atorvastatin 10 mg QD via oral tablet for the entire duration of the study. Double-blind atorvastatin is to be added to the regimen for participants not achieving LDL-C target (≤100 mg/dL; 2.59 mmol/L). The maximum possible total daily dose of atorvastatin received in this group is 80 mg (10 mg open label plus 70 mg double blind).
  Interventions: Drug: Atorvastatin; Drug: Placebo for Atorvastatin
- Ezetimibe + Atorvastatin (Experimental): Participants receive double-blind ezetimibe 10 mg QD via oral tablet PLUS open-label atorvastatin 10 mg QD via oral tablet for the entire duration of the study. Double-blind atorvastatin is to be added to the regimen for participants not achieving LDL-C target (≤100 mg/dL; 2.59 mmol/L). The maximum possible total daily dose of atorvastatin received in this group is 40 mg (10 mg open label plus 30 mg double blind).
  Interventions: Drug: Atorvastatin; Drug: Ezetimibe; Drug: Placebo for Ezetimibe; Drug: Placebo for Atorvastatin

INTERVENTIONS:
Drug: Atorvastatin — Atorvastatin administered orally QD as 10 mg tablets.
  Other Names: LIPITOR®; SCH 412387; MK-9396
Drug: Ezetimibe — Ezetimibe administered orally QD as 10 mg tablets
  Other Names: ZETIA®; SCH 058235; MK-0653
  Arms: Ezetimibe + Atorvastatin
Drug: Placebo for Ezetimibe — Single placebo tablet administered orally QD
  Arms: Ezetimibe + Atorvastatin
Drug: Placebo for Atorvastatin — Single placebo tablet administered orally QD

SUMMARY:
The overall objective is to evaluate the efficacy and safety of ezetimibe (SCH 058235/MK-0653) 10 mg administered daily in conjunction with atorvastatin in participants with Heterozygous Familial Hypercholesterolemia (HeFH) or in participants with coronary heart disease (CHD) or multiple cardiovascular risk factors (≥2 risk factors) and primary hypercholesterolemia not controlled by a starting dose (10 mg/day) of atorvastatin.

The primary hypothesis is that the coadministration of ezetimibe 10 mg/day with atorvastatin therapy will result in a significantly greater proportion of participants achieving target low-density lipoprotein cholesterol (LDL-C) (≤100 mg/dL) when compared to the atorvastatin administered alone.

ELIGIBILITY:
Inclusion Criteria:

* Primary hypercholesterolemic participants with known coronary heart disease (CHD) or multiple risk factors for CHD (≥2) not meeting the target low-density-lipoprotein cholesterol (LDL-C) of ≤100 mg/dL (2.59 mmol/L), with plasma LDL-C ≥130 mg/dL (3.37 mmol/L) and plasma triglycerides (TG) ≤350 mg/dL (3.99 mmol/L) while on starting-dose (10 mg) atorvastatin at least 4 weeks before initial qualifying lipid determination.
* Participants with heterozygous familial hypercholesterolemia (HeFH) not meeting the target LDL-C of ≤100 mg/dL (2.59 mmol/L), with plasma LDL-C ≥130 mg/dL (3.37 mmol/L) and plasma TG ≤350 mg/dL (3.99 mmol/L) while on starting-dose (10 mg) atorvastatin for at least 4 weeks before initial lipid qualifying determination. HeFH is defined by: a) genetic testing; or b) LDL-C >190 mg/dL (4.9 mmol/L) and at least one of the following: (1) xanthomata in first or second degree relative; (2) family history of myocardial infarction under age 60 years in a first degree relative or family history of myocardial infarction under age 50 years in a second degree relative; (3) family history of total cholesterol (TC) >290 mg/dL (>7.5 mmol/L) in a first or second degree relative.
* All women must have a negative pregnancy test prior to study entry. Women of child-bearing potential must agree to practice an effective barrier method of birth control for the duration of the study, as well as for 1 month following study completion.
* Postmenopausal women who are receiving postmenopausal hormonal therapy or raloxifene must be maintained on a stable estrogen replacement therapy (ERT), estrogen/progestin hormone replacement therapy (HRT) or raloxifene regimen during the study period.
* Participants must be willing to observe the National Cholesterol Education Program (NCEP) Step I diet as determined by a Ratio of Ingested Saturated fat and Cholesterol to Calories (RISCC) score not greater than 24 throughout this study. Ability to complete diet diaries needs to be demonstrated.

Exclusion Criteria:

* Individuals with a history of mental instability, drug/alcohol abuse within the past 5 years or individuals who have been treated or are being treated for severe psychiatric illness which in the opinion of the Investigator, may interfere with optimal participation in the study.
* Underlying disease likely to limit life span to less than 1 year.
* Participants who have previously been randomized in any of the studies evaluating ezetimibe.
* Participants with known hypersensitivity or any contraindication to atorvastatin
* Pregnant or lactating women.
* Participants with congestive heart failure New York Heart Association (NYHA) Class III or IV.
* Participants with uncontrolled cardiac arrhythmias
* Participants with myocardial infarction, coronary bypass surgery or angioplasty within 3 months of study entry.
* Participants with unstable or severe peripheral artery disease within 3 months of study entry.
* Participants with unstable angina pectoris.
* Participants with disorders of the hematologic, digestive or central nervous systems including cerebrovascular disease and degenerative disease that would limit study evaluation or participation.
* Participants with uncontrolled (as determined by hemoglobin A1c [HbA1c]) or newly diagnosed (within 1 month of study entry) diabetes mellitus.
* Participants with uncontrolled endocrine or metabolic disease known to influence serum lipids or lipoproteins. Clinically euthyroid participants on replacement doses of thyroid hormone are eligible for enrollment.
* Participants with known impairment of renal function (creatinine >2.0 mg/dL), dysproteinemia, nephrotic syndrome or other renal disease (24-hour urinary protein 3+ or 1 gram).
* Participants with active or chronic hepatobiliary or hepatic disease (participants with aspartate aminotransferase (AST) or alanine aminotransferase (ALT) >2 times the upper limit of the central laboratory reference range [ULN] will be excluded).
* Participants who are known to be human immunodeficiency virus (HIV) positive.
* Participants with known coagulopathy (prothrombin time [PT] or partial thromboplastin time [PTT] at Visit 2 >1.25 times control).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 621 (Actual)
Dates: Start 2000-04-24 (Actual); Primary Completion 2001-11-16 (Actual); Study Completion 2001-11-16 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants Achieving Target Low-Density-Lipoprotein Cholesterol (LDL-C) Levels of ≤100 mg/dL | Week 14
  The percentage of participants achieving the target low-density-lipoprotein cholesterol (LDL-C) levels (≤100 mg/dL [2.59 mmol/L]) as determined from blood samples following a standard ultracentrifugation/precipitation procedure (β-quantification).
Percentage of Participants With an Adverse Event | 14 weeks (Up to 16 weeks)
  An adverse event (AE) is defined as any physical or clinical change or disease reported by a participant or observed by the investigator or member of the staff at any time during the study, regardless of potential relationship to study treatment, and included onset or discovery of new illness and exacerbation of any pre-existing condition.
Percentage of Participants Who Discontinued the Study due to an Adverse Event | 14 weeks (Up to 16 weeks)
  An adverse event (AE) is defined as any physical or clinical change or disease reported by a participant or observed by the investigator or member of the staff at any time during the study, regardless of potential relationship to study treatment, and included onset or discovery of new illness and exacerbation of any pre-existing condition.

SECONDARY OUTCOMES:
Percentage of Participants Achieving Target LDL-C level (≤100 mg/dL) | Week 4
  The percentage of participants achieving the target low-density-lipoprotein cholesterol (LDL-C) levels (≤100 mg/dL [2.59 mmol/L]) as determined from blood samples following a standard ultracentrifugation/precipitation procedure (β-quantification).
Mean Percent Change from Baseline in Direct LDL-C | Baseline and Week 4
  Participants are to have their direct LDL-C levels assessed at baseline and after 4 weeks of study drug administration. The change from baseline will be calculated.
Mean Percent Changes from Baseline for Calculated LDL-C | Baseline and Week 4
  Participants are to have their calculated LDL-C levels assessed at baseline and after 4 weeks of study drug administration. The change from baseline will be calculated.
Mean Percent Changes from Baseline for Total Cholesterol (TC) | Baseline and Week 4
  Participants are to have their TC levels assessed at baseline and after 4 weeks of study drug administration. The change from baseline will be calculated.
Mean Percent Changes from Baseline for Triglycerides (TG) | Baseline and Week 4
  Participants are to have their TG levels assessed at baseline and after 4 weeks of study drug administration. The change from baseline will be calculated.
Mean Percent Changes from Baseline for High-Density-Lipoprotein Cholesterol (HDL-C) | Baseline and Week 4
  Participants hare to have their HDL-C levels assessed at baseline and after 4 weeks of study drug administration. The change from baseline will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Stein E, Stender S, Mata P, Sager P, Ponsonnet D, Melani L, Lipka L, Suresh R, Maccubbin D, Veltri E; Ezetimibe Study Group. Achieving lipoprotein goals in patients at high risk with severe hypercholesterolemia: efficacy and safety of ezetimibe co-administered with atorvastatin. Am Heart J. 2004 Sep;148(3):447-55. doi: 10.1016/j.ahj.2004.03.052. PMID 15389231